CLINICAL TRIAL: NCT06493240
Title: Neoadjuvant Long-course Chemoradiotherapy Followed by PD-1 Monoclonal Antibody for Locally Advanced Mid-low Rectal Cancer
Brief Title: Neoadjuvant Long-course Chemoradiotherapy Followed by Immunotherapy for Locally Advanced Mid-low Rectal Cancer
Acronym: NLCCRIT-LARC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shen Zhanlong, Department of Gastroenterological Surgery, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023PHB222; Z220014 (Other Grant/Funding Number: Beijing Municipal Natural Science Foundation)
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Locally Advanced Rectal Cancer; PD-1 inhibition; neoadjuvant therapy
MeSH Terms: interventions — Radiation; spartalizumab; sintilimab

STUDY DESIGN:
Masking Description: Masking is not practically possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nCRT+PD-1 (Experimental): Long-course chemoradiation followed by PD-1 inhibition (Sintilimab 200mg, 3 times, 2-week interval) starting on Day 15 after completion of radiation therapy. TME surgery is scheduled in 6 weeks after completion of radiation.
  Interventions: Radiation: radiation; Drug: PD-1 Monoclonal Antibody; Procedure: TME surgery

INTERVENTIONS:
Radiation: radiation — 45 Gy radiation dose in 25 fractions to the pelvis
Drug: PD-1 Monoclonal Antibody — 200mg Sintilimab after radiation (3 times, 2-week interval)
  Other Names: Sintilimab
Procedure: TME surgery — TME surgery for 6~8 weeks after radiation
  Other Names: radical proctectomy

SUMMARY:
The purpose of this study was to evaluate the effect of capecitabine-based long-term radiotherapy followed by 3 cycles Sintilimab (PD-1 inhibitor) in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
Investigator designed a single-arm, open-label, phase II trial and the purpose of this study is to observe and evaluate the efficacy and safety of capecitabine-based long-term radiotherapy followed by 3 cycles Sintilimab (PD-1 inhibitor) for locally advanced rectal cancer.Participants will accept capecitabine-based long-term radiotherapy(50.4Gy radiation) followed by 200mg Sintilimab each time for 3 times, with 2-week intervals. The primary endpoint is pCR rate, and secondary endpoints include sphincter-preserving rate, adverse event rates.

ELIGIBILITY:
Inclusion Criteria:

* aged 18~75
* ECOG score 0~2
* biopsy diagnosed rectal adenocarcinoma, distal margin within 10cm to anal verge
* no distant metastasis, staged II/III (T4b excluded) by MRI
* maximum diameter of rectal cancer lesion≥10mm according to baseline CT or MR
* willing and able to comply with study protocol
* consent to the use of blood and tissue specimens for study
* no history of previous anti-tumor treatment (e.g. radiation, chemo, immuno, bio, herbal, etc.)
* no disorders/diseases of immune system (e.g. systemic lupus erythematosus, rheumatoid arthritis, systemic vasculitis, scleroderma, pemphigus, dermatomyositis, mixed connective tissue disease, autoimmune hemolytic anemia, hyperthyroidism/hypothyroidism, ulcerative colitis, autoimmune hemolytic anemia, HIV infection, etc.)
* no significant dysfunction of major viscera (e.g. heart, lung, liver, kidney, etc.)
* no jaundice or gastrointestinal obstruction
* no acute/ongoing infection
* no significant irregularities in blood routine test and biochemical test results, particular requirements include: neutrophils≥1.5×109/L, HGB≥80g/L, platelet≥100×109/L, serum creatinine≤1.5×ULN, total bilirubin≤1.5×ULN, ALT、AST≤2.5×ULN
* no social or mental disorder
* for women of child-bearing age, a negative result of serological pregnancy test is required, and effective contraception measures from inclusion till 60 days after the last dose of study drug is required

Exclusion Criteria:

* multiple cancers, or with concomitant malignant tumors besides rectal cancer
* having received any anti-cancer treatment (surgery, drugs, etc.) in the past 5 years
* history of recent major surgery
* with condition that affects the absorption of capecitabine via gastrointestinal tract (e.g. inability to swallow, nausea, vomiting, chronic diarrhea, etc.)
* with uncontrolled, severe, concomitant diseases of any sort
* allergic to any of the ingredients under study
* estimated survival ≤ 5 years due to any reason
* preparing for or having previously received organ or bone marrow transplant
* having received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to inclusion
* for patients with history of disorder of central nervous system, investigator discretion is required as to whether the clinical severity prevents the signing of informed consent or affects the patient or oral medication compliance
* with other conditions/issues that may affect the study results or cause the study treatment to be terminated halfway (e.g. alcoholism, drug abuse, etc.)
* pregnant or lactating women, or women intending on conception during treatment period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
pCR rate | within 1 week after surgery
  pathological complete response rate

SECONDARY OUTCOMES:
sphincter preserving rate | instantly after surgery
  proportion of patients with preserved anal sphincter
immune-related adverse event rate | from commencing of PD-1 inhibition to the 30th day after surgery
  adverse event rate that is deemed to be associated with PD-1 inhibition
treatment-related adverse event rate | from commencing of treatment to the 30th day after surgery
  adverse event rate that is deemed to be associated with all treatments
incidence rate of surgical complications | within 30 days after surgery
  incidence rate of surgical complications within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhanlong Zhanlong, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Export of individual patient data is a sensitive issue according to current Chinese laws